CLINICAL TRIAL: NCT04773496
Title: Normative Data for Static and Dynamic Posturography (NeuroCom EQUITEST and BALANCE MASTER) in Subjects Older Than 79yrs
Acronym: EQUIOLD
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 24C402
Record Dates: First submitted 2021-02-19; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Equilibrium; Disorder, Labyrinth; Aging
Keywords: normative data; postural balance; posturography; EquiTest®; Sensory Organization Test; aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Balance evaluation: patient's balance is evaluated with instrumental posturography
  Interventions: Diagnostic Test: instrumental description of the subject's center of gravity (COG) sway

INTERVENTIONS:
Diagnostic Test: instrumental description of the subject's center of gravity (COG) sway — qualitative and quantitative analysis of the balance function through the description of the center of gravity (COG) sway

SUMMARY:
Ageing is known to increase the risk of fall and posturographic stabilometry, both static and dynamic, are useful tools to assess postural stability. To our knowledge, no published normative data for a healthy elderly population are available.

DETAILED DESCRIPTION:
The risk of fall rise with ageing and is huge after 85yrs becoming one of the major problems associated with aging.

The computed dynamic posturographic EquiTest® System and Smart BalanceMaster by NeuroCom® International, Inc, Clackamas, OR, USA) provide a qualitative and quantitative analysis of the balance function through the description of the subject's center of gravity (COG) sway.

Sensory Organization Test and Sensory Analysis norms are provided for age groups (20-59; 60-69; 70-79) up to 79yrs, whilst they lack in the international literature for subjects 80+yrs, nonetheless being necessary in the understanding of balance performance from a quantitative point of view.

Subjects 80+yrs are evaluated with EquiTest® System and Smart BalanceMaster to provide mean values and normative data.

In order to assess the reliability of the instrumental evaluation was repeated (T1) two weeks later (±2 days).

ELIGIBILITY:
Inclusion Criteria:

* Age older than 79 years
* Free gait, without aids, for at least 50 mt
* Cognitive skills allowing the providing of valid informed consent and the understanding of the instructions during clinical and instrumental evaluations

Exclusion Criteria:

* Pathologies affecting Central Nervous System (i.e., cerebrovascular, neurodegenerative, Alzheimer Disease, Parkinson disease, etc) or vestibulum
* Previous traumatic brain injury and/or coma lasting more than 24 hrs and occurred within last 20 years
* Impairment affecting the Peripheral Nervous System i.e., pallesthesia <4/8
* Hip or knee joint replacement within the last 10 years
* Surgeries or pathologies affecting the lower limbs or the spine
* Pain, acute or chronic
* Use, within the last 12 hours, of painkillers or drugs interfering with Central Nervous System or balance

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Subjects 80+yrs were enrolled from the general healthy Italian population.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Normative Data for Sensory Organization Test with EquiTest® System in subjects aged 80yrs and over | instrumental evaluation is performed at enrollment;
  Center of gravity sway during posture is evaluated through computed dynamic posturographic EquiTest® System.

SECONDARY OUTCOMES:
Normative Data for Motor Control Test and Adaptation Test with EquiTest® System in subjects aged 80yrs and over | instrumental evaluation is performed at enrollment
  Motor responses during perturbations posture are evaluated through computed dynamic posturographic EquiTest® .
Normative Data for dynamic tests with Smart BalanceMaster® System in subjects aged 80yrs and over | instrumental evaluation is performed at enrollment
  Center of gravity sway during posture is evaluated through computed dynamic posturographic Smart BalanceMaster® System.
Reliability of the measures (measures stability) | Instrumental evaluation is repeated two weeks after enrollment
  To verify that the instrument yields the same results over multiple trials a second evaluation is performed a second time

CONTACTS AND LOCATIONS:
Overall Officials: LAURA PERUCCA, MD, Study Chair — ISTITUTO AUXOLOGICO ITALIANO IRCCS - UNIVERSITA DEGLI STUDI DI MILANO
Locations (2):
- Italy (2):
  - Istituto Auxologico Italiano, Irccs, Milan, Lombardy
  - Fondazione Irccs Ospedale Maggiore Policlinico, Milan

IPD SHARING:
Plan to Share IPD: Yes